CLINICAL TRIAL: NCT04305431
Title: Exploring a Dietary Behavior Intervention in African-Americans at Risk for Cardiovascular Disease: A Community Acceptability and Feasibility Study
Brief Title: Dietary Behavior Intervention in African Americans at Risk for Cardiovascular Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 200036; 20-CC-0036
Record Dates: First submitted 2020-03-11; First posted 2020-03-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12-05

CONDITIONS: Diet; Cooking
Keywords: Diabetes; Heart Disease; Dietary Behavior; Nutrition
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1/All Subjects (Experimental): Second phase participants
  Interventions: Behavioral: Cooking Intervention

INTERVENTIONS:
Behavioral: Cooking Intervention — 90-minute culinary education sessions.

SUMMARY:
Background:

The risk of heart disease among African Americans is still common despite a greater understanding of the disease and better approaches to managing it. Healthy cooking and eating patterns can help reduce the risk of heart disease. But things like access to grocery stores and knowledge of good nutrition can affect these healthy patterns. Researchers want to see if community-based programs can help.

Objective:

To learn about the cooking behaviors of African American adults at risk for heart disease. Also, to see if a community-based cooking intervention will affect home-cooking behaviors.

Eligibility:

African American adults 18 and older who live in Wards 7 and 8 of Washington, D.C., and have at least one self-reported risk factor for heart disease

Design:

Phase I participants will complete a survey. It asks about their medical history, lifestyle, stress level, and eating habits. They will take part in a focus group. During this, they will talk about what they eat and what foods are available to them. Participation lasts 1 day for 3 hours at Pennsylvania Avenue Baptist Church in Washington, D.C.

Phase II participants will go to shared cooking events at Pennsylvania Avenue Baptist Church. These will be held once a week for 6 weeks. They will be led by a trained chef. Participants will visit the NIH Clinical Center 3 times. Transportation will be provided if they need it. They will have physical exams and have blood drawn. They will be interviewed and complete questionnaires. A dietician will review the food they eat. An occupational therapist will assess their cooking skills. They will keep a daily cooking journal. Participation lasts 18 weeks.

DETAILED DESCRIPTION:
Study Description: Explore feasibility measures, facilitators and barriers related to cooking and cooking frequency among an AA adult population at risk for CVD following participation in a cooking intervention.

Objectives:

First Phase Primary Objective:

Identify facilitators and barriers to cooking frequency and assess feasibility of a cooking intervention among AA adults living in a food desert community.

Assess feasibility of a cooking intervention among AA adults living in a food desert community.

First Phase Secondary Objectives:

Explore the relationship between cooking frequency, facilitators, and barriers with individual, social environment and built environment factors, as suggested from qualitative research and cooking intervention studies.

Second Phase Primary Objectives:

Identify facilitators and barriers to cooking, and cooking frequency among AA adults living in a food desert community who participate in a cooking intervention.

Determine feasibility measures of the intervention associated with cooking frequency, facilitators, or barriers for participants who participate in a cooking intervention.

Second Phase Secondary Objectives:

Explore the relationship between feasibility measures, cooking frequency, facilitators and barriers with individual factors, social environment and built environment factors related to cooking at home as a result of participating in a cooking intervention

Explore the relationship between feasibility measures, cooking frequency, facilitators and barriers to dietary quality, as determined by evaluation of food dietary records, Mediterranean Diet Score, Healthy Eating Index scores for participants who participate in a cooking intervention.

Explore the relationship between feasibility measures, cooking frequency, facilitators and barriers with CVD biomarkers, as measured by CVD related laboratory studies, and anthropometric measurements.

Endpoints:

Primary Endpoint:

Identify and measure barriers, facilitators, cooking frequency, cooking skills in AA participants: in context of feasibility risibility measures for the cooking intervention.

Secondary Endpoints:

Explore and measure diet quality and CVD biomarkers.

ELIGIBILITY:
* FIRST PHASE:

A sample of AA adults (n= 20) living in Wards 7 or 8 of Washington, D.C. will be recruited for this phase.

INCLUSION CRITERIA:

English-speaking

Self-identified AA adults (defined as age greater than or equal to 18)

Live in Wards 7 or 8 in Washington, D.C.

At least one self-reported risk factor for CV disease known by participant or told to participant by a clinician within the last 12 months. Specific risk factors are:

* overweight or obese (self-reported height and weight compute to BMI if needed greater than or equal to 25)
* elevated waist to hip ratio
* elevated cholesterol
* clinical hypertension or prehypertension
* prediabetes
* elevated fasting glucose level on laboratory report
* current smoker or prior (within the past 12 months) smoker.

EXCLUSION CRITERIA:

Under the age of 18

Do not live in Wards 7 or 8 in Washington, D.C.

No risk factors for CVD

Or adults not of AA descent (self-identified)

Non-English speaking

SECOND PHASE:

A sample of AA adults (n= 35) living in Wards 7 or 8 of Washington, D.C. will be recruited for this phase.

INCLUSION CRITERIA:

English-speaking

Self-identified AA adults (defined as age greater than or equal to 18)

Who live in Wards 7 or 8 in Washington, D.C.

At least one self-reported risk factor for CV disease known by participant or told to participant by a clinician within the last 12 months. Specific risk factors are:

* overweight or obese (self-reported height and weight compute to BMI if needed >= 25)
* elevated waist to hip ratio
* elevated cholesterol
* clinical hypertension or prehypertension
* prediabetes
* elevated fasting glucose level on laboratory report
* current smoker or prior (within the past 12 months) smoker.

Not pregnant at the time of screening and enrollment.*

Willing to not attend or enroll in another cooking/culinary education program or class during participation in this study

Not enrolled currently or in the prior 12 months (at time of recruitment) in another ongoing cooking/culinary education program or class

EXCLUSION CRITERIA:

AAs who are not age greater than or equal to 18

AA Adults not living in Wards 7 or 8 in Washington, D.C.

AA Adults living in the same household as another participant

AA adults without at least one risk factor for CVD

Or adults not of AA descent

Non-English speaking

Those enrolled currently or in the prior 12 months at time of recruitment in another ongoing cooking/culinary education program

Those not willing to not attend or enroll in another cooking/culinary education program or class during participation in this study

* If individuals become pregnant during their participation, they can continue to participate if they want to. The pregnant participant will not undergo DEXA scanning procedure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2026-12-19 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Measures | 26 weeks
  Recruitment and retention/attrition Attendance/Dosage Participant burden Implementation- treatment fidelity; measures of home cooking behavior
Facilitators and Barriers | 26 weeks
  Cooking diaries Cooking Self-Efficacy Scale D.C. CHOC Cooking Survey Cooking and Food Provisioning Action Scale AMPS (cooking skill) score

SECONDARY OUTCOMES:
Second Phase Secondary Outcome | 18 weeks
  Social Network Index HPLP-II Perceived Stress Scale MESA Neighborhood Healthy Food Availability Scale Perceptions of Neighborhood Food Retail Outlets Neighborhood Satisfaction Food purchasing practices Self-rated Health Pittsburgh Sleep Quality Assessment International Physical Activity Questionnaire-Short Form Food Away from Home Purchasing Frequency Family Meals Eaten Together Grocery receipts CVD related laboratory biomarkers Antropometric mesurements

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Farmer, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Farmer N, Tuason RT, Kazmi N, Flynn S, Mitchell V, Middleton K, Cox R, Franklin K, Gordon T, Baginski A, Wallen GR. Going virtual during the COVID-19 pandemic: adaptation of a mixed-methods dietary behavior study within a community-based participatory research study of African-American adults at risk for cardiovascular disease. BMC Med Res Methodol. 2022 Dec 22;22(1):330. doi: 10.1186/s12874-022-01806-3. PMID 36550396
- [Derived] Farmer N, Powell-Wiley TM, Middleton KR, Roberson B, Flynn S, Brooks AT, Kazmi N, Mitchell V, Collins B, Hingst R, Swan L, Yang S, Kakar S, Harlan T, Wallen GR. A community feasibility study of a cooking behavior intervention in African-American adults at risk for cardiovascular disease: DC COOKS (DC Community Organizing for Optimal culinary Knowledge Study) with Heart. Pilot Feasibility Stud. 2020 Oct 19;6:158. doi: 10.1186/s40814-020-00697-9. eCollection 2020. PMID 33088581
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-CC-0036.html